CLINICAL TRIAL: NCT00677495
Title: Usefulness of Gluten-free Diet in Gluten-genetically Predisposed Subjects Positive to Intestinal-mucosa Anti-transglutaminase Antibodies
Brief Title: Gluten-free Diet in Gluten-genetically Predisposed Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Collaborators: University of Trieste (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Luca Ronfani, MD, IRCCS Burlo Garofolo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC 25/07
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Genetic Predisposition to Disease; Celiac Disease
Keywords: Gluten-free diet; Celiac Disease; Genetic predisposition; Phage display library; Autoimmune diseases
MeSH Terms: conditions — Genetic Predisposition to Disease; Celiac Disease; Autoimmune Diseases | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gluten-free diet (Experimental): Gluten-free diet
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — Gluten-free diet

SUMMARY:
Undetected or untreated CD may cause severe complications later in life, such as autoimmune disorders.

It is recommended for subjects with autoimmune diseases or at risk for CD to be screened for CD and to repeat serological screening about every three years to detect cases of clinically silent, late-onset CD.

Celiac disease (CD) auto-antibodies against tissue transglutaminase (anti-tTG) are produced in the intestinal mucosa even when not measurable in serum. By using the phage display libraries technique it is possible to investigate in vivo (intestinal biopsy) early antibody responses in autoimmune disease. In particularly, this technique demonstrated that the humoral response against tissue transglutaminase occurs at the intestinal mucosal level, and that the human VH5 gene is the commonly used variable region by the celiac patients to build the anti-tTG. The intestinal mucosa production of IgA anti-tTG could be important in the diagnostic work-up of early-stage CD, when mucosal histology is not yet diagnostic.

The investigators propose to 1) first degree relatives of CD patients, 2) subjects with autoimmune disease, 3) symptomatic subjects (genetically predisposed to gluten intolerance) tested negative for CD related autoantibodies and with apparently normal intestinal mucosa a prospective study to uncover early-stage of gluten intolerance by measuring the mucosal VH5 restricted gene family anti-tTG clones in two biopsies: before and after one year of gluten free-diet (GFD).

Aims of this clinical trial are:

1. to measure by means of phage display libraries the gluten dependent humoral immune response (anti-tTG) of the intestinal mucosa in subjects with high risk of untreated CD, without CD-related intestinal lesions.
2. to demonstrate the mucosal gluten-dependent immune response before and after 12 months of gluten-free diet
3. to demonstrate that dietary intervention might modify the clinical condition (e.g improvements of the gastrointestinal complaints or extra-gastrointestinal symptoms) of the enrolled patients and the improvement of the intestinal inflammation with the disappearance of the mucosal anti-tTG.
4. to evaluate the specificity of the double staining technique for detecting IgA antitransglutaminase mucosal deposit with the phage display antibodies assay

DETAILED DESCRIPTION:
Celiac disease (CD) is an autoimmune enteropathy triggered by ingestion of gluten in genetically susceptible subjects and is one of the most frequently occurring, treatable, lifelong disorders. In this disease we recognize the trigger (gluten), the genetic factor (HLA DQ2/8), the auto-antigen (the tissue-transglutaminase enzyme) and the auto-antibodies (IgA-IgG anti-transglutaminase) which are produced by the intestinal mucosa B lymphocytes (Gastroenterology 2000;119:234, J Immunol 2001;166:4170). Undetected or untreated, CD may cause more severe complications later in life, such as autoimmune disorders. Clear evidence exists of gluten-related autoimmunity in genetically predisposed patients (presence of the HLA DQ2/8). It has been shown that autoimmune disorders involving organs other than intestine (such as pancreas, cerebellum, liver, skin) could develop in unrecognized and/or untreated celiac subjects because of a persistent exposure to gluten. Presently, the additional risk for autoimmune diseases is estimated at 1.1% for each year without diagnosis (Gastroenterology 1999;117:297). Furthermore, when on a diet containing gluten, some CD patients produced organ-specific auto-antibodies (GAD, ICA, TPO, anti-Purkinje cells, cardiac auto-antibodies) which were not CD related and which disappeared after 6 to 12 months of gluten-free diet (J Pediatr 2000;137:263; Lancet 1996;347:369; Circulation 2002;105:2611). Bearing these data in mind, an early diagnosis of CD might have prevented some CD patients from developing an autoimmune disease such as type 1 diabetes or thyroiditis. In view of these observations, it is recommended for subjects with autoimmune diseases or at risk for CD to be screened for CD and to repeat serological screening about every three years to detect cases of clinically silent, late-onset CD. In other words, there are gluten-genetically predisposed subjects (tested positive for HLA DQ2/8) - testing negative for serum anti-tTG - that become antibody-positive later in life. The tTG-targeted antibodies bound locally to tissue transglutaminase may be present in diseased organs before they become detectable in the circulation, thus accessible for serological testing. The intestinal mucosa in the early phases is characterized by normal villi including a normal number of intraepithelial lymphocytes. The process of mucosal deterioration may take years or even decades (Am J Gastroenterol 2000;95:463) and a long follow-up without treatment may sometimes be harmful. Symptoms are not related solely to villous atrophy, and many proven early celiac disease cases had suffered from gluten-dependent gastrointestinal symptoms even before the villous atrophy developed (Gut 2006;55:133, Scand J Gastroenterol 2005;40:564, Gut 2004;53:641, Scand J Gastroenterol 1998;33:944, Acta Paediatr 1995;84:1252, Gastroenterology 1993;104:1263).

By using the phage display libraries technique it is possible to investigate in vivo (intestinal biopsy) early antibody responses in autoimmune disease. In particularly, this technique demonstrated that the humoral response against tissue transglutaminase occurs at the intestinal mucosal level, and that the human VH5 gene is the commonly used variable region by the immune system of CD-patients to build the anti-tTG. This means that phage display libraries technique is able to measure the specificity of the autoimmune response against the tissue transglutaminase enzyme and perhaps against others auto-antigens (GAD, ICA, TPO, cardiac-antigens) in the CD patients. Phage display libraries allow us to measure the specific auto-antibodies at the production site, also in patients testing negative for anti-tTG in the serum and allow us to identify early CD patients before their seroconversion and the deterioration of their jejunal mucosa. Therefore, the intestinal mucosa production of IgA anti-tTG could be important in the diagnostic work-up of early-stage CD, when mucosal histology is not yet diagnostic.

The investigators propose to first degree relatives of CD patients with or without symptoms and to subjects with autoimmune disease tested negative for serum anti-tTG but positive for CD related HLA DQ2 or DQ8 a prospective study to uncover early-stage of gluten intolerance by measuring the mucosal VH5 restricted gene family anti-tTG clones in two biopsies: before and after one year of gluten free-diet (GFD). Symptomatic subjects genetically predisposed to gluten intolerance, tested negative for CD related autoantibodies and with apparently normal intestinal mucosa, were also enrolled for detecting the deposits of IgA transglutaminase at intestinal level and, after one year of gluten free diet, and to evaluate the clinical modifications.

Aims of this clinical trial are:

1. to measure by means of phage display libraries the gluten dependent humoral immune response (anti-tTG) of the intestinal mucosa in subjects with high risk of untreated CD, without CD-related intestinal lesions.
2. to demonstrate the mucosal gluten-dependent immune response before and after 12 months of gluten-free diet.
3. to demonstrate that dietary intervention might modify the clinical condition (e.g improvements of the gastrointestinal complaints or extra-gastrointestinal symptoms) of the enrolled patients and the improvement of the intestinal inflammation with the disappearance of the mucosal anti-tTG.
4. to evaluate the specificity of the double staining technique for detecting IgA antitransglutaminase mucosal deposit with the phage display antibodies assay

ELIGIBILITY:
Inclusion Criteria:

* first degree relatives of CD patients
* subjects with autoimmune disease tested negative for serum anti-tTG but positive for CD related HLA DQ2 or DQ8
* symptomatic subjects (genetically predisposed to gluten intolerance) tested negative for CD related autoantibodies and with apparently normal intestinal mucosa.

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Intestinal mucosal gluten-dependent immune response before and after a gluten-free diet | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Ziberna, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy; Serena Vatta, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy; Stefano Martelossi, MD, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy; Roberto Marzari, Principal Investigator — University of Trieste; Fiorella Florian, Principal Investigator — University of Trieste; Vincenzo Villanacci, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia; Daniele Sblattero, Principal Investigator — Department of Medical Sciences, University of Eastern Pidmont, Novara, Italy; Alessandro Ventura, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Tarcisio Not, MD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Not T, Ziberna F, Vatta S, Quaglia S, Martelossi S, Villanacci V, Marzari R, Florian F, Vecchiet M, Sulic AM, Ferrara F, Bradbury A, Sblattero D, Ventura A. Cryptic genetic gluten intolerance revealed by intestinal antitransglutaminase antibodies and response to gluten-free diet. Gut. 2011 Nov;60(11):1487-93. doi: 10.1136/gut.2010.232900. Epub 2011 Apr 6. PMID 21471568
- [Derived] De Leo L, Quaglia S, Ziberna F, Vatta S, Martelossi S, Maschio M, Not T. Serum anti-tissue transglutaminase antibodies detected during febrile illness may not be produced by the intestinal mucosa. J Pediatr. 2015 Mar;166(3):761-3. doi: 10.1016/j.jpeds.2014.12.005. PMID 25722272